CLINICAL TRIAL: NCT02433717
Title: A Study on the Efficacy, Pharmacokinetics and Adverse Effects of Paliperidone ER
Brief Title: A Pharmacokinetic Study of Paliperidone ER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201501049MINC
Record Dates: First submitted 2015-04-16; First posted 2015-05-05 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; pharmacogenetics; pharmacokinetics; event-related potentials; paliperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paliperidone ER (Experimental): Six-week paliperidone ER
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — Fixed dose (9 mg/day) of paliperidone ER will be given in the first two weeks of trial (from day 1 to day 14). Since the third week (day 15), the dosage can be adjusted in the range of 6 to 12 mg per day.
  Other Names: Invega

SUMMARY:
Background Paliperidone is an active metabolite of risperidone, both of which are antipsychotic agents for treatment of schizophrenia and related psychotic disorders. Pharmacogenetic studies have revealed that the efficacy and side effects of antipsychotic agents are related to polymorphisms of specific genes, however, there are just a few related studies on paliperidone. The current study aims to evaluate whether pharmacogenetic markers related to risperidone and genetic markers associated with schizophrenia have effects on the clinical effectiveness of paliperidone treatment. The study also uses changes of event-related potentials (ERP) as indices for clinical efficacy.

Methods It is a prospective, open-label, non-randomized and uncontrolled clinical trial to study the efficacy and side effects of 6-week paliperidone ER treatment for patients with schizophrenia or schizoaffective disorder. The first three weeks of treatment has to be inpatient treatment. In the first two weeks, participants will take 9 mg paliperidone ER daily. Then the dose of paliperidone can be adjusted to within the range of 6-12 mg per day. Efficacy indicators include symptom severity, global functioning, and ERP. Side effect indicators include common side effect evaluate, extrapyramidal symptoms, metabolic profiles, hormonal change, and bone metabolism indices. Participants will also receive examinations for blood drug concentration, genetic polymorphisms, and epigenetic markers.

DETAILED DESCRIPTION:
A. Background Schizophrenia is a heterogeneous disorder whose pathophysiology is not yet understood clearly. The treatment of schizophrenia remains suboptimal. Take risperidone for example, response rate of a patient is around only 60% to 80%. The second-generation or atypical antipsychotics are widely used. Apart from dopamine D2 receptor, they also target on 5-HT2 receptors and receptors of other neurotransmission systems. However, these second-generation antipsychotics still result in other common side effects. Therefore, finding predictors for clinical efficacy and side effect profile is a necessary task. Up to date, several genetic and non-genetic factors have been suggested related to the efficacy and side effects of antipsychotics. Noteworthy, pharmacokinetics as indicated by the temporal change of antipsychotics blood levels is usually overlooked. It might be a contributing factor why results from pharmacogenetic studies were usually difficult to be replicated.

Paliperidone (9-hydroxy-risperidone) is an active metabolite of the second-generation antipsychotics risperidone. Pharmacogenetic studies have found polymorphisms of some genes to be related to blood risperidone concentration, side effects and treatment response. Comparing to risperidone, paliperidone has less metabolic side effects, probable faster occurrence of efficacy, and better tolerance for subjects with hepatic insufficiency. Further, paliperidone is more sensitive to P-glycoprotein. There are just a few pharmacogenetic studies on paliperidone and P-glycoprotein. Therefore, one aim of this proposed study is to examine the pharmacogenetic effects on paliperidone extended release (paliperidone ER) for acute treatment of schizophrenia and schizoaffective disorder. The electrophysiological abnormalities as measured by event-related potentials (ERP) are characteristics features of several neuropsychological disorders. For schizophrenia, deficits in mismatch negativity, P50, and auditory steady state response have been frequently reported. Therefore, besides from clinical improvements, the investigators are also interested whether paliperidone treatment can alter the deficits in mismatch negativity, P50, and ASSR.

B. Study aims

1. To study the association of candidate genes, which are related to pharmacodynamics and pharmacokinetics of risperidone, with paliperidone pharmacokinetics and clinical response
2. To evaluate the impact of pharmacodynamics on the efficacy (including ERP change and cognitive function) and side effects of paliperidone ER for acute treatment of schizophrenia
3. To evaluate whether the paliperidone pharmacodynamics is related to the metabolic, hormonal, and bone turnover profiles
4. To evaluate whether paliperidone ER treatment will influence epigenetic markers
5. To evaluate whether paliperidone ER treatment will influence event-related potentials and performance in neurocognitive tests

C. Study design It is a 6-week, prospective, open-label, uncontrolled and non-randomized trial of paliperidone ER for patients with schizophrenia or schizoaffective disorder in an acute episode. A total of 40 subjects will be recruited.

D. Protocol overview:

For at least the first three weeks, participants should receive inpatient treatment in the acute psychiatry ward (03W2) in National Taiwan University Hospital. Medication compliance, efficacy of treatment and side effects will be monitored and evaluated by the psychiatrists who are the principle investigator or sub-investigators of this study.

1. Dosage of titration of paliperidone ER:

   Fixed dose (9 mg/day) of paliperidone ER will be given in the first two weeks of trial (from day 1 to day 14). Since the third week (day 15), the dosage can be adjusted in the range of 6 to 12 mg per day.
2. Medication regulation:

   1. Antipsychotics other than paliperidone ER are not allowed.
   2. For benzodiazepines and sedatives/hypnotics: only lorazepam up to 4 mg per day is allowed to management medication withdrawal, side effects or symptoms.
   3. Anticholinergic agents: for management of extrapyramidal symptoms only biperiden up to 6 mg/day or trihexyphenidyl up to 15 mg/day is allowed.
3. Measurements 3-1. Clinical evaluation on day 0, day 4, day 7, day14, day 28, and day 42:

   1. Efficacy evaluation: positive and Negative Syndrome Scale (PANSS), Personal and Social Performance Scale (PSP), Clinical Global Impression-Severity (CGI-S)
   2. Side effect evaluation: Drug-Induced Extrapyramidal Symptom Scale (DIEPSS), and Udvalg for Kliniske Undersogelser (UKU) Side Effect Rating Scale; any new-onset adverse conditions or worsening of the original conditions will be recorded as side effects and be managed promptly.
   3. Body weight. 3-2. Blood sampling on day 0 (40 ml), day 14 (15 ml) and day 42 (40 ml):

   <!-- -->

   1. Blood paliperidone concentration and pharmacodynamics of risperidone and paliperidone on day 0, day 14, and day 42.
   2. Blood biochemistry study (AC sugar, uric acid, cholesterol, triglyceride, HDL-cholesterol, leptin, adiponectin, prolactin) on day 0, day 14, and day 42.
   3. Bone turnover markers (serum alkaline phosphatase, calcium, phosphate bone-specific alkaline phosphatase, intact osteocalcin), and hormonal markers (oestradiol, progesterone, LH, FSH and testosterone) on day 0 and day 42.
   4. DNA sample for genetic markers on day 0: 1236C/T of the ABCB1 gene, Ser9Gly of the DRD3 gene, Ser311Cys of the DRD2 gene, 267T/C of the 5HTR6 gene, 102T/C of the 5HTR2A gene, 995G/A of the 5HTR2C gene, dinucleotide repeat (GT)n of the BDNF gene, val108/158Met of the COMT gene, and polymorphisms of the RGS4 gene.
   5. Epigenetic markers on day 0 and day 42. 3-3. Urinary examination for bone turnover markers on day 0 and day 42: urinary deoxypyridinoline cross-links and urinary C-terminal telopeptide fragment of type I collagen 3-4. Electrocardiogram on day 0 and day 42. 3-5. Event-related potential experiments on day 0 and day 42: Participants will receive experiments of mismatch negativity, P50 and auditory steady state response 3-6. Neurocognitive tests on day 0 and day 42: Participants will receive Continuous Performance Test (CPT), Wisconsin Card Sorting Test (WCST), Trail-A test, Trail-B test, verbal fluency test, and selected subtests from Wechsler Adult Intelligence Test-III (Digit Span and Arithmetic).

D. Conditions when a subject drop-out from the trial

1. Whenever a subject withdraws the informed consent.
2. Whenever a serious treatment-emergent adverse event happens.
3. Whenever the treating psychiatrists or the principle investigator judge early dropout necessary for a subject, considering the risks and benefits clinically.
4. Whenever a subject violates the trial protocol to a significant degree, as judged by the treating psychiatrists or the principle investigator.

E. Conditions when the trial will be stopped Since paliperidone ER has been approved for the treatment of schizophrenia by the Food and Drug Administration and the daily dose is within the recommended range, this trial will be terminated or suspended under the following situations: (a) order from the Research Ethics Committee to terminate or suspend the clinical trial; (b) order from the Central Competent Health Authority to terminate or suspend the clinical trial; (c) when paliperidone ER becoming unavailable in the National Taiwan University Hospital.

F. Trial medications Paliperidone Extended-Release Tablets (Invega): 9 mg/tab, 3 mg/tab

G. Data collection and statistical analysis

Since the current study is an open-labeled and single-arm trial, it is not aimed to prove the efficacy of paliperidone for treatment of schizophrenia. Instead, it is aimed to evaluate whether pharmacodynamics factors are related to the clinical response of paliperidone treatment. The variables of clinical response are defined as:

1. Primary efficacy variable: response rate (the ratio of subjects who respond to paliperidone treatment).

   Response to paliperidone treatment is calculated as [(PANSSevaluation - PANSSbaseline)/ (PANSSbaseline -30)]*100%
2. Secondary efficacy variables: PSP, CGI-S, ERPs and neurocognitive tests
3. Side effect variables: DIEPSS, UKU side effect scales, body weight, blood chemistry markers, metabolic markers, hormonal markers, and bone turnover markers

Response rate and other efficacy variables were analyzed with last observation carried forward and intention-to-treat principles. Response rate will be calculated on day 4, 7, 14, 28 and 42, and the impact of pharmacodynamics and genetic effects will be analyzed accordingly. Demographic data, blood paliperidone concentration, and the aforementioned variables will be compared between responder group and non-responder group on last visit (Pearson χ2 test or Fisher exact test will be used to compare categorical variables; independent t test will be used for continuous variables). The secondary efficacy and side effect variables on day 0 (before treatment) and day 42 (after treatment) will be compared with paired t-test. Relationship of the change of the aforementioned variables with blood paliperidone concentration will be examined by Pearson's correlation coefficient test or Spearman's correlation coefficient test. Multiple linear regression analysis will be applied for adjustments of covariates.

The genotyping quality will be checked by Hardy-Weinberg equilibrium tests. Association of the allelic effects of the genetic markers with clinical response and other outcome variables will be analyzed by using PLINK version 1.07 19. Other statistical analyses will be performed by using SAS®9.4 Software (SAS Institute Inc., USA). A p-value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion criteria:

* 20-65 years old
* With DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Being hospitalized in an acute psychiatric ward
* Scoring at least 60 according to the Positive and Negative Syndrome Scale (PANSS)
* Having not received long-acting injectable antipsychotics in the past 6 months
* Having no major physical disorders or significant abnormalities in laboratory studies

Exclusion criteria:

* Having abused illicit substances in the past 6 months
* Having physical disorders that may influence the absorption, metabolism, or excretion of paliperidone ER
* With substantial suicidal or violence risk
* Being pregnant or lactating, or with high probability of getting pregnant
* With other significant central nervous system abnormalities
* With other significant unstable or incurable physical illnesses
* Having ever taken clozapine in the past 3 months
* Having ever taken paliperidone ER within 30 days before eligibility evaluation
* History of allergy to paliperidone ER or risperidone
* Without the competence to sign the informed consent
* Hearing impairments

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics factor on response rate | day 42
  Whether the concentration of blood paliperidone is related to the clinical response rate on day 42. Clinical response is defined as achieving 50% or more improvement in terms of PANSS total score:
  [(PANSS at evaluation - PANSS at baseline)/ (PANSS at baseline - 30)]*100% ≥ 50%
Pharmacogenetic factor on response rate: ABCB1 | day 42
  Whether 1236C/T of the ABCB1 gene is associated with the clinical response rate on day 42.
Pharmacogenetic factor on response rate: DRD3 | day 42
  Whether Ser9Gly of the DRD3 gene is associated with the clinical response rate on day 42.
Pharmacogenetic factor on response rate: DRD2 | day 42
  Whether Ser311Cys of the DRD2 gene is associated with the clinical response rate on day 42.
Pharmacogenetic factor on response rate: 5HTR6 | day 42
  Whether 267T/C of the 5HTR6 gene is associated with the clinical response rate on day 42.
Pharmacogenetic factor on response rate: 5HTR2A | day 42
  Whether 102T/C of the 5HTR2A gene is associated with the clinical response rate on day 42.
Pharmacogenetic factor on response rate: 5HTR2C | day 42
  Whether 995G/A of the 5HTR2C gene is associated with the clinical response rate on day 42.
Pharmacogenetic factor on response rate: BDNF | day 42
  Whether dinucleotide repeat (GT)n of the BDNF gene is associated with the clinical response rate on day 42.
Pharmacogenetic factor on response rate: COMT | day 42
  Whether val108/158Met of the COMT gene is associated with the clinical response rate on day 42.
Pharmacogenetic factor on response rate: RGS4 | day 42
  Whether polymorphisms of RGS4 gene is associated with the clinical response rate on day 42.

SECONDARY OUTCOMES:
Change in person and social function | day 4, day 7, day14, day 28, and day 42
  Measured by Personal and Social Performance Scale (PSP)
Change in global impression of the patient | day 4, day 7, day14, day 28, and day 42
  Measured by Clinical Global Impression-Severity (CGI-S) 2. Side effect variables: DIEPSS, UKU side effect scales, body weight, blood chemistry markers, metabolic markers, hormonal markers, and bone turnover markers
Change in mismatch negativity | day 42
  Mismatch negativity is an event-related potential measurement
Change in P50 | day 42
  P50 is an event-related potential measurement
Change in auditory steady state response | day 42
  Auditory steady state response is an event-related potential measurement
Change in attention as measured by Continuous Performance Test (CPT) | day 42
  CPT is a neurocognitive test
Change in executive function as measured by Wisconsin Card Sorting Test (WCST) | day 42
  WCST is a neurocognitive test
Change in performance on Trail-A test | day 42
  Trail-A test is a neurocognitive test
Change in performance on Trail-B test | day 42
  Trail-B test is a neurocognitive test
Change in performance on verbal fluency test | day 42
  Verbal fluency test is a neurocognitive test
Change in performance on Digit Span | day 42
  Digit Span is a subtest of Wechsler Adult Intelligence Test-III
Change in performance on Arithmetic | day 42
  Arithmetic is a subtest of Wechsler Adult Intelligence Test-III
Pharmacodynamics and pharmacogenetics factors on response rate | day 4, day 7, day14, day 28
  Clinical response are defined as 50% or more improvement in terms of PANSS total score:
  [(PANSS at evaluation - PANSS at baseline)/ (PANSS at baseline - 30)]*100% ≥ 50%
Severity of extrapyramidal symptoms | day 4, day 7, day14, day 28, day 42
  Severity of extrapyramidal symptoms is measured by Drug-Induced Extrapyramidal Symptom Scale (DIEPSS)
Severity of side effects | day 4, day 7, day14, day 28, day 42
  Severity of side effects is measured by Udvalg for Kliniske Undersogelser (UKU) Side Effect Rating Scale
Effects on blood glucose level | day 14 and day 42
  AC sugar
Effects on blood cholesterol level | day 14 and day 42
Effects on blood triglyceride level | day 14 and day 42
Effects on blood HDL-cholesterol level | day 14 and day 42
Effects on blood prolactin level | day 14 and day 42
Effects on blood leptin level | day 14 and day 42
Effects on adiponectin level | day 14 and day 42
Effects on blood alkaline phosphatase level | day 42
Effects on blood calcium level | day 42
Effects on blood phosphate level | day 42
Effects on blood bone-specific alkaline phosphatase level | day 42
Effects on blood intact osteocalcin level | day 42
Effects on blood oestradiol level | day 42
Effects on blood progesterone level | day 42
Effects on blood LH level | day 42
Effects on blood FSH level | day 42
Effects on blood testosterone level | day 42
Effects on blood uric acid level | day 14 and day 42

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ting Lin, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Taiwan
  - Department of Psychiatry, National Taiwan University Hospital, Taipei, Test2